CLINICAL TRIAL: NCT05919641
Title: LIVELUNG - Impact of CGA on QoL, Overall Survival and the Need for Admission in Patients Diagnosed With Localized NSCLC Treated With SBRT - a National Randomized Study
Brief Title: LIVELUNG - Impact of CGA in Patients Diagnosed With Localized NSCLC Treated With SBRT
Acronym: LIVELUNG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kirkelund Bentsen, Dr.med., Odense University Hospital
Other Study IDs: LIVELUNG
Record Dates: First submitted 2023-06-12; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer; Stereotactic Body Radiotherapy; Comprehensive Geriatric Assessment
Keywords: NSCLC; SBRT; CGA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- +CGA: Patients randomised to undergo a Comprehensive Geriatric Assessment (CGA)
  Interventions: Other: Comprehensive Geriatric Assessment
- -CGA: Patients not randomised to undergo a Comprehensive Geriatric Assessment (CGA)

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Comprehensive geriatric assessment (CGA) is defined as a multidisciplinary diagnostic and treatment process that identifies medical, psychosocial, and functional capabilities of an older adult in order to develop a coordinated plan to maximize overall health with aging.
  Groups: +CGA

SUMMARY:
Older patients with non-small cell lung cancer (NSCLC) treated with stereotactic body radiation therapy (SBRT) often die from other causes than lung cancer due to age-related comorbidities. This national randomized study will include 130 patients throughout 5 Danish cancer centres and investigate if a comprehensive geriatric intervention (CGA) when added upfront to SBRT for patients with localized NSCLC will have an impact on quality of life (QoL), overall survival, physical functionality and unplanned hospital admissions.

If an upfront CGA improves patients' general health status, this study could lead to implementation of a CGA in standard clinical practice as well as further research on older patients receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically or histologically proven non-small cell lung cancer
* Stage T1-3N0M0
* ≥ 70 years old
* In a multidisciplinary setting the patient is considered medically inoperable, too frail for operation due to age and/or comorbidity or that the patient refuse surgery and therefore candidate for SBRT.

Exclusion Criteria:

* Missing histology/cytology
* Another current malignancy
* Higher staging at treatment planning
* Not able to provide informed consent
* Do not speak or understand Danish

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients, able to provide informed consent, aged ≥70 diagnosed with T1-3N0M0 NSCLC considered medically inoperable at a multidisciplinary setting and therefore candidates for SBRT. 130 patients will be included in a period of 24 months.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EQ-5D) | 12 months
  Questionnaire with 5 dimensions each with 5 (1-5) levels representing the health status of the patient and the patients self-rated health status on a scale from 0-100 (EQ VAS). The score of the 5 dimensions can be converted into a single index value 0-1 with higher values indicating poorer health status.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  The time from treatment to death, regardless of disease recurrence
Quality of Life (EQ-5D) | 3 months
  Questionnaire with 5 dimensions each with 5 (1-5) levels representing the health status of the patient and the patients self-rated health status on a scale from 0-100 (EQ VAS). The score of the 5 dimensions can be converted into a single index value 0-1 with higher values indicating poorer health status.
Quality of Life (EQ-5D) | 6 months
  Questionnaire with 5 dimensions each with 5 (1-5) levels representing the health status of the patient and the patients self-rated health status on a scale from 0-100 (EQ VAS). The score of the 5 dimensions can be converted into a single index value 0-1 with higher values indicating poorer health status.
Quality of Life (EQ-5D) | 9 months
  Questionnaire with 5 dimensions each with 5 (1-5) levels representing the health status of the patient and the patients self-rated health status on a scale from 0-100 (EQ VAS). The score of the 5 dimensions can be converted into a single index value 0-1 with higher values indicating poorer health status.
Hand-grip strength | 12 months
  Hand-grip strength measured in kilo using a JAMAR hand dynamometer
Timed-up-and-go (TUG) | 12 months
  TUG consists of timing (seconds) a patient getting up from a chair from the sitting to the bipedal position, walking three meters, turning, returning, and sitting on the chair again
Chair-stand-test (CST) | 12 months
  The CST involves recording the number of "stands" from a chair a person can complete in 30 seconds
Unplanned Admissions | 12 months
  Time to first unplanned admission

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Bentsen, Dr. med, Principal Investigator — Department of Oncology, Odense University Hospital, Denmark
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No